CLINICAL TRIAL: NCT00146328
Title: A Long Term Open Label Rollover Trial Assessing the Safety and Tolerability of Combination Tipranavir and Ritonavir Use in HIV-1 Infected Subjects
Brief Title: Rollover Trial Safety and Tolerability of Combination Tipranavir and Ritonavir Use in HIV 1 Infected Subjects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.17
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir

ARMS (3):
- Group 1 (Experimental): Patients With Varying Degrees of Tipranavir Treatment Experience
  Interventions: Drug: Tipranavir
- Group 2 (Experimental): Highly Tipranavir Treatment Experienced Patients
  Interventions: Drug: Tipranavir
- Group 3 (Experimental): Tipranavir Treatment Naive Patients
  Interventions: Drug: Tipranavir

INTERVENTIONS:
Drug: Tipranavir

SUMMARY:
The objective of this study is to determine the long term safety and tolerability of multiple oral doses of tipranavir (Aptivus) and ritonavir with a focus on the long term safety of the development dose (500 mg tipranavir/200 mg ritonavir BID) when administered with other antiretroviral medications.

ELIGIBILITY:
INCLUSION CRITERIA

1. Ability and willingness to give written informed consent in accordance with institutional and federal guidelines and to comply with the investigational nature of the study and the related requirements.
2. All subjects must have successfully completed participation in a combination tipranavir/ritonavir trial or have confirmed virologic failure in the 1182.12 or 1182.48 trials and are not able to obtain TPV by prescription. Successful completion of participation is defined as conclusion of required subject-weeks on assigned dosing (trial specific) and completion of required visits.
3. Male and female subjects 18 years and over.
4. Presence of Human Immunodeficiency Virus 1 (HIV-1) infection as documented by any licensed Enzyme Linked immunosorbent Assay (ELISA) test kit and confirmed by Western Blot, or HIV-1 culture, or HIV-1 antigen, or plasma HIV 1 Ribonucleic Acid (RNA) or a second antibody test by a method other than ELISA at any time prior to study entry.
5. Adherence to previous tipranavir/ritonavir dosing protocol and adherence to visit requirements of previous protocol (as assessed by principal investigator).
6. Acceptable screening laboratory values that indicate adequate baseline organ function. Laboratory values are considered to be acceptable if the following apply:

   * Total Cholesterol ≤400 mg/dl (<Common Toxicity Criteria (CTC) Grade 2).
   * Total Triglycerides ≤750 mg/dl (<Division of AIDS (DAIDS) Grade 2).
   * Alanine aminotransferase (ALT) ≤3.0x upper limit of normal (ULN) and Aspartate aminotransferase (AST) ≤2.5x ULN (<DAIDS Grade 1).
   * Any Grade Gamma Glutamyl transpeptidase(GGT) is acceptable.
   * Any Grade creatinine kinase is acceptable as long as there is no concurrent myopathy.
   * All other laboratory test values ≤DAIDS Grade 1.

EXCLUSION CRITERIA

1. Female subjects who are of reproductive potential who:

   * Have a positive serum beta human chorionic gonadotropin (B HCG) at Screening/Enrollment Visit.
   * Are not willing to use a reliable method of barrier contraception (such as diaphragm or condoms).
   * Are breast-feeding.
2. Subjects who are actively using injection drugs or other substance abuse (such as extensive alcohol or narcotic use) which is considered by the investigator to be a significant impairment to health and to protocol adherence.
3. Any medical condition(s) which, in the opinion of the investigator, would interfere with the subject's ability to participate in or adhere to the requirements of this protocol.
4. History of any illness or drug allergy which, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering tipranavir/ritonavir to the subject.
5. Active use of any of the following:

   * Investigational HIV-1 vaccines.
   * Any new investigational antiretroviral agent that was not approved for use in the patients prior tipranavir trial.
   * Medications excluded during the trial period (see Section 4.2).
   * Herbal medications (e.g., St. John's Wort).
6. Active HIV-related or non HIV-related illness that may be negatively affected by use of tipranavir/ritonavir as determined by the investigator.

   If a subject must temporarily discontinue tipranavir/ritonavir at the recommendation of the investigator (at the completion of the previous tipranavir trial), then the subject may enroll in 1182.17 once the clinical illness has resolved, and after approval from the Boehringer Ingelheim Clinical Monitor or Local Clinical Monitor.
7. Clinically significant liver disease in the 90 days prior to baseline visit, regardless of baseline AST and/or ALT values.
8. Hypersensitivity to tipranavir or ritonavir.
9. Voluntary discontinuation of antiretroviral therapy (including tipranavir/ritonavir) for more than seven days from completion of previous tipranavir trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 997 (Actual)
Dates: Start 2001-04; Primary Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (233):
- United States (86):
  - 1182.17.39 MDS Pharma Services, Phoenix, Arizona
  - 1182.17.75 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1182.17.89 Boehringer Ingelheim Investigational Site, Berkeley, California
  - 1182.17.60 Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - 1182.17.106 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1182.17.15 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1182.17.40 Tower ID Medical, Los Angeles, California
  - 1182.17.46 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1182.17.47 University of Southern California, Los Angeles, California
  - 1182.17.73 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1182.17.114 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1182.17.128 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1182.17.37 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1182.17.58 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1182.17.96 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1182.17.87 Boehringer Ingelheim Investigational Site, Norwalk, Connecticut
  - 1182.17.112 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1182.17.43 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1182.17.65 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1182.17.126 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1182.17.8 Boehringer Ingelheim Investigational Site, Fort Myers, Florida
  - 1182.17.131 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1182.17.22 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1182.17.64 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1182.17.129 Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - 1182.17.51 Boehringer Ingelheim Investigational Site, South Miami, Florida
  - 1182.17.125 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1182.17.132 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1182.17.76 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1182.17.52 Boehringer Ingelheim Investigational Site, Vero Beach, Florida
  - 1182.17.77 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1182.17.69 Boehringer Ingelheim Investigational Site, Macon, Georgia
  - 1182.17.136 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1182.17.70 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1182.17.36 Boehringer Ingelheim Investigational Site, Evanston, Illinois
  - 1182.17.1 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1182.17.32 University of Kansas School of Medicine - Wichita, Wichita, Kansas
  - 1182.17.102 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 1182.17.21 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1182.17.30 Boehringer Ingelheim Investigational Site, Portland, Maine
  - 1182.17.67 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1182.17.86 Boehringer Ingelheim Investigational Site, Bethesda, Maryland
  - 1182.17.111 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1182.17.63 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1182.17.74 Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - 1182.17.4 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 1182.17.115 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 1182.17.6 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 1182.17.62 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1182.17.59 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1182.17.118 Early Intervention Program (EIP) Clinic, Camden, New Jersey
  - 1182.17.93 Boehringer Ingelheim Investigational Site, East Orange, New Jersey
  - 1182.17.24 Hackensack University Medical Center, Hackensack, New Jersey
  - 1182.17.34 ID Care, Inc., Hillsborough, New Jersey
  - 1182.17.50 Boehringer Ingelheim Investigational Site, Santa Fe, New Mexico
  - 1182.17.79 Boehringer Ingelheim Investigational Site, Albany, New York
  - 1182.17.103 Boehringer Ingelheim Investigational Site, Mount Vernon, New York
  - 1182.17.105 Pollari Medical Group, New York, New York
  - 1182.17.130 Boehringer Ingelheim Investigational Site, New York, New York
  - 1182.17.3 Division of Infectious Diseases, New York, New York
  - 1182.17.42 Beth Israel Medical Center, New York, New York
  - 1182.17.5 Boehringer Ingelheim Investigational Site, New York, New York
  - 1182.17.7 Boehringer Ingelheim Investigational Site, New York, New York
  - 1182.17.94 Boehringer Ingelheim Investigational Site, New York, New York
  - 1182.17.135 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1182.17.31 Boehringer Ingelheim Investigational Site, Stony Brook, New York
  - 1182.17.53 Boehringer Ingelheim Investigational Site, Durham, North Carolina
  - 1182.17.54 Boehringer Ingelheim Investigational Site, Huntersville, North Carolina
  - 1182.17.134 Summa Health System, Akron, Ohio
  - 1182.17.95 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1182.17.26 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1182.17.9 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1182.17.110 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1182.17.99 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1182.17.23 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 1182.17.11 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1182.17.18 Vanderbilt AIDS Clinical Trials Center, Nashville, Tennessee
  - 1182.17.116 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1182.17.142 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1182.17.16 Nelson-Tebedo Clinic, Dallas, Texas
  - 1182.17.122 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1182.17.68 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1182.17.97 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1182.17.10 Boehringer Ingelheim Investigational Site, Annandale, Virginia
  - 1182.17.92 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 1182.17.100 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin
- Argentina (6):
  - 1182.17.5401 Fundacion Huesped, Capital Federal
  - 1182.17.5402 Funcei, Capital Federal
  - 1182.17.5403 consultorio externo "PETS", Capital Federal
  - 1182.17.5404 Infectología, Capital Federal
  - 1182.17.5405 Dpto. de Enfermedades infecciosas (Pabellón 22), Capital Federal
  - 1182.17.5406 Pabellón de Clínicas 2° Piso, Capital Federal
- Australia (7):
  - 1182.17.401 St. Vincent's Hospital, Darlinghurst, New South Wales
  - 1182.17.402 Taylor Square Private Clinic, Darlinghurst, New South Wales
  - 1182.17.405 AIDS Research Initiative, Darlinghurst, New South Wales
  - 1182.17.407 Holdsworth House General Practice, Darlinghurst, New South Wales
  - 1182.17.408 407 Doctors Pty Ltd., Darlinghurst, New South Wales
  - 1182.17.403 Albion Street Clinic, Surry Hills, New South Wales
  - 1182.17.404 Alfred Hospital, Melbourne, Victoria
- 1182.17.4301 Boehringer Ingelheim Investigational Site, Vienna, Austria
- Belgium (5):
  - 1182.17.3209 Instituut Tropische Geneeskunde, Antwerp
  - 1182.17.3201 Boehringer Ingelheim Investigational Site, Brussels
  - 1182.17.3202 Boehringer Ingelheim Investigational Site, Brussels
  - 1182.17.3207 Boehringer Ingelheim Investigational Site, Ghent
  - 1182.17.3210 Centre Hospitalier de Luxembourg, Luxembourg
- Brazil (11):
  - 1182.17.5511 Universidade Federal da Bahia, Canela - Salvador - BA
  - 1182.17.5508 I.I. Emilio Ribas, Cerqueira César, São Paulo - SP
  - 1182.17.5509 (Unidade de Testes Terapêuticos), Cidade Nova - Rio de Janeiro - RJ
  - 1182.17.5502 Farmácia do Instituto de Pesquisa Evandro Chagas, Manguinhos - Rio de Janeiro - RJ
  - 1182.17.5505 Instituto A-Z de Pesquisa e Ensino da PUC, Mercês - Curitiba - PR
  - 1182.17.5507 Hospital Geral de Nova Iguaçu - Ministério da Saúde, Nova Iguaçu - Rio de Janeiro - RJ
  - 1182.17.5501 Hospital Dia, Sacoma - São Paulo - SP
  - 1182.17.5503 Instituto de Infectologia Emílio Ribas, São Paulo - SP
  - 1182.17.5504 Enfermaria de MI, São Paulo - SP
  - 1182.17.5510 Casa de AIDS, São Paulo, SP
  - 1182.17.5506 Centro de Referência e Treinamento - DST/AIDS, Vila Mariana, Sao Paulo - SP
- Canada (11):
  - 1182.17.902 Downtown Infectious Diseases Clinic, Vancouver, British Columbia
  - 1182.17.913 McMaster University Medical Centre, Hamilton, Ontario
  - 1182.17.901 Division of Infectious Diseases, Ottawa, Ontario
  - 1182.17.905 Canadian Immunodeficiency Research Collaborative Inc., Toronto, Ontario
  - 1182.17.906 Infectious Diseases & HIV - St. Michael's Hospital, Toronto, Ontario
  - 1182.17.907 University Health Network - Toronto General Hospital, Toronto, Ontario
  - 1182.17.910 Sunnybrook & Women's College Health Science Centre, Toronto, Ontario
  - 1182.17.914 Montreal General Hospital - McGill University Health Centre, Monteal, Quebec
  - 1182.17.903 Montreal Chest Institute, McGill University Health Centre, Montreal, Quebec
  - 1182.17.904 Clinique Medicale Du Quartier Latin, Montreal, Quebec
  - 1182.17.915 Clinique medicale l'Actuel, Montreal, Quebec
- Denmark (4):
  - 1182.17.4505 Boehringer Ingelheim Investigational Site, Aarhus N
  - 1182.17.4501 Boehringer Ingelheim Investigational Site, Copenhagen Ø
  - 1182.17.4502 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1182.17.4504 Boehringer Ingelheim Investigational Site, Odense
- France (22):
  - 1182.17.33011 Hôpital Pellegrin, Bordeaux
  - 1182.17.33019 Hôpital Saint André, Bordeaux
  - 1182.17.33020 Hôpital Côte de Nacre, Caen
  - 1182.17.33007 Hôpital Antoine Beclere, Clamart
  - 1182.17.33008 Hôpital de l'Hôtel Dieu, Lyon
  - 1182.17.33023 Hôpital Edouard Herriot, Lyon
  - 1182.17.33012 Hôpital de la Conception, Marseille
  - 1182.17.33013 Hôpital Sainte Marguerite, Marseille
  - 1182.17.00336 Hôpital Hôtel Dieu, Nantes
  - 1182.17.33010 Hôpital de l'Archet, Nice
  - 1182.17.00331 Hôpital Tenon, Paris
  - 1182.17.00333 Hôpital Saint Louis, Paris
  - 1182.17.00334 Hôpital de la Pitié Salpêtrière, Paris
  - 1182.17.00335 Hôpital Bichat Claude Bernard, Paris
  - 1182.17.33014 Hôpital Saint Antoine, Paris
  - 1182.17.33022 Hôpital Européen Georges Pompidou, Paris
  - 1182.17.33024 Groupe Hospitalier Cochin, Paris
  - 1182.17.33018 Hôpital de Pontchaillou, Rennes
  - 1182.17.33016 Hôpital Civil, Strasbourg
  - 1182.17.00332 Hôpital du Chalucet, Toulon
  - 1182.17.33017 Hôpital Brabois Adultes, Vandœuvre-lès-Nancy
  - 1182.17.33021 Hôpital Paul Brousse, Villejuif
- Germany (24):
  - 1182.17.4911 Arzt für Innere Medizin, Aachen
  - 1182.17.4901 Epimed GmbH c/o, Berlin
  - 1182.17.4902 Charite, Campus Virchow-Klinikum, Berlin
  - 1182.17.4918 Rheinische Friedrich-Wilhelm-Universität, Bonn
  - 1182.17.4905 Universitätsklinik Köln, Cologne
  - 1182.17.4926 Internist, Cologne
  - 1182.17.4906 ID-Ambulanz Klinikum Dortmund, Dortmund
  - 1182.17.4912 Universitätsklinikum Düsseldorf, Düsseldorf
  - 1182.17.4914 Arzt für Innere Medizin, Düsseldorf
  - 1182.17.4908 Universitätskliniken Erlangen, Erlangen
  - 1182.17.4904 Universitätsklinikum Essen, Essen
  - 1182.17.4924 Klinikum der J. W.-Goethe-Universität, Frankfurt am Main
  - 1182.17.4928 Facharzt für Innere Medizin/Rheumatologie, Freiburg im Breisgau
  - 1182.17.4930 Universitätsklinikum Freiburg, Freiburg/Breisgau
  - 1182.17.4916 Medizinisches Versorgungszentrum Hamburg, Hamburg
  - 1182.17.4929 Universitätsklinikum Eppendorf, Hamburg
  - 1182.17.4931 IPM Study Center GmbH, Hamburg
  - 1182.17.4920 Abteilung Klinische Immunologie, Hanover
  - 1182.17.4909 Universitätsklinikum Heidelberg, Heidelberg
  - 1182.17.4923 Facharzt für Innere Medizin,, Mannheim
  - 1182.17.4907 Medizinische Poliklinik, München
  - 1182.17.4910 MUC Research GmbH, München
  - 1182.17.4915 Klinium Natruper Holz, Osnabrück
  - 1182.17.4921 Arzt für Allgemeinmedizin, Stuttgart
- Greece (7):
  - 1182.17.3001 Boehringer Ingelheim Investigational Site, Athens
  - 1182.17.3002 Boehringer Ingelheim Investigational Site, Athens
  - 1182.17.3003 Boehringer Ingelheim Investigational Site, Athens
  - 1182.17.3004 Boehringer Ingelheim Investigational Site, Athens
  - 1182.17.3007 Boehringer Ingelheim Investigational Site, Athens
  - 1182.17.3010 Boehringer Ingelheim Investigational Site, Pátrai
  - 1182.17.3009 Boehringer Ingelheim Investigational Site, Thessaloniki
- Italy (17):
  - 1182.17.0409 Ospedale Santa Maria Annunziata, Antella (fi)
  - 1182.17.0413 Ospedale di Circolo di Busto, Busto Arsizio (va)
  - 1182.17.0384 Azienda Ospedaliera Arcispedale S. Anna, Ferrara
  - 1182.17.0397 Ospedale San Martino, Genova
  - 1182.17.0412 S.C. Malattie Infettive, Genova
  - 1182.17.0411 Presidio Ospedaliero "A. Manzoni", Lecco
  - 1182.17.0389 Reparto Malattie Infettive, Macerata
  - 1182.17.0393 Fondazione Centro S. Raffaele del Monte Tabor, Milan
  - 1182.17.0386 Policlinico Universitario, Modena
  - 1182.17.0388 Ospedale A. Cotugno, Napoli
  - 1182.17.0385 IRCCS Policlinico San Matteo, Pavia
  - 1182.17.0394 IRCCS Policlinico San Matteo, Pavia
  - 1182.17.0395 Azienda Policlinico Umberto I, Roma
  - 1182.17.0419 I Cattedra Malattie Infettive, Roma
  - 1182.17.0387 Ospedale Amedeo di Savoia, Torino
  - 1182.17.0398 Ospedale Amedeo di Savoia, Torino
  - 1182.17.0415 U.O.A. Malattie Infettive B, Torino
- Mexico (3):
  - 1182.17.5201 Centro Médico La Raza IMSS, Col. La Raza, Mexico
  - 1182.17.5203 Hospital Civil Nuevo de Guadalajara, Guadalajara
  - 1182.17.5206 Centro Medico San Vicente, Monterrey, N.l., Mexico
- Netherlands (4):
  - 1182.17.3101 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1182.17.3108 Boehringer Ingelheim Investigational Site, Groningen
  - 1182.17.3105 Boehringer Ingelheim Investigational Site, Nijmegen
  - 1182.17.202 Boehringer Ingelheim Investigational Site, Rotterdam
- 1182.17.3502 Hospital Condes Castro Guimarães, Cascais, Portugal
- Spain (11):
  - 1182.17.705 Hospital Germans Trias i Pujol, Badalona
  - 1182.17.701 Hospital Clínico y Provincial de Barcelona, Barcelona
  - 1182.17.703 Hospital 12 de Octubre, Madrid
  - 1182.17.704 Hospital Ramón y Cajal., Madrid
  - 1182.17.710 Hospital Gregorio Maranon, Madrid
  - 1182.17.712 Hospital Clínico San Carlos, Madrid
  - 1182.17.717 Hospital Clínico Universitario Vírgen de la Victoria, Málaga
  - 1182.17.713 Hospital Universitario Vírgen del Rocío, Seville
  - 1182.17.714 Hospital General Universitario de Valencia, Valencia
  - 1182.17.720 Hospital La Fe, Valencia
  - 1182.17.718 Complejo Hospitalario Xeral - Cíes, Vigo
- Switzerland (4):
  - 1182.17.4101 DIM / Abteilung für Infektiologie, Basel
  - 1182.17.4104 Département de médicine interne Div. Des maladies infectieus, Geneva
  - 1182.17.4103 DIM / Abteilung für Infektiologie, Sankt Gallen
  - 1182.17.4102 Departement für Innere Medizin, Zurich
- United Kingdom (9):
  - 1182.17.4405 Boehringer Ingelheim Investigational Site, Brighton
  - 1182.17.4411 Boehringer Ingelheim Investigational Site, Liverpool
  - 1182.17.4404 Boehringer Ingelheim Investigational Site, London
  - 1182.17.4406 Boehringer Ingelheim Investigational Site, London
  - 1182.17.4408 Boehringer Ingelheim Investigational Site, London
  - 1182.17.4409 Boehringer Ingelheim Investigational Site, London
  - 1182.17.4414 Boehringer Ingelheim Investigational Site, London
  - 1182.17.4418 Boehringer Ingelheim Investigational Site, London
  - 1182.17.4407, Portsmouth

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (Patients With Varying Degrees of Treatment Experience: Group 1: TPV/r patients who rolled over from Trials 1182.2, 1182.4, 1182.6, 1182.52 (NCT00275444, NCT00034866), 1182.12 (NCT00054717) and 1182.48 (NCT00144170). A total of 291 patients were categorized into Group 1.
- Group 2 (Highly Treatment Experienced Patients): Group 2: Patients from 1182.51 (NCT00056641) who rolled over into 1182.17. A total of 255 patients were categorized into Group 2.
- Group 3 (Tipranavir naïve Patients): Group 3: PI comparator arm patients from 1182.4, 1182.12 (NCT00054717) and 1182.48 (NCT00144170) who virologically failed and who then rolled into 1182.17. A total of 449 patients were categorized into Group 3.
Period: Overall Study
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Started | 291 | 255 | 449
Completed | 150 | 101 | 158
Not Completed | 141 | 154 | 291
Not completed — Adverse Event | 39 | 48 | 79
Not completed — Protocol Violation | 11 | 6 | 12
Not completed — Lost to Follow-up | 7 | 4 | 7
Not completed — Withdrawal by Subject | 16 | 16 | 22
Not completed — Virologic Failure/lack of efficacy | 54 | 72 | 142
Not completed — Trial ended/site closed | 8 | 2 | 19
Not completed — Patient decision to end | 0 | 1 | 6
Not completed — Enroll into other trial | 2 | 4 | 2
Not completed — Death | 0 | 1 | 1
Not completed — Moved | 2 | 0 | 0
Not completed — Interaction with other medication | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1 (Patients With Varying Degrees of Treatment Experience: A total of 995 patients who entered 1182.17 from a 'core' TPV/r trial were treated with TPV/r and were included in the integrated database. Of the 995 patients from 241 sites in 19 countries worldwide, 291 patients were categorized into Group 1. Group 1: TPV/r patients who rolled over from Trials 1182.2, 1182.4, 1182.6, 1182.52, 1182.12 and 1182.48.
- Group 2 (Highly Treatment Experienced Patients): A total of 995 patients who entered 1182.17 from a 'core' TPV/r trial were treated with TPV/r and were included in the integrated database. Of the 995 patients from 241 sites in 19 countries worldwide, 255 patients were categorized into Group 2. Group 2: Patients from 1182.51 who rolled over into 1182.17.
- Group 3 (Tipranavir naïve Patients): A total of 995 patients who entered 1182.17 from a 'core' TPV/r trial were treated with TPV/r and were included in the integrated database. Of the 995 patients from 241 sites in 19 countries worldwide, 449 patients were categorized into Group 3. Group 3: PI comparator arm patients from 1182.4, 1182.12 and 1182.48 who virologically failed and who then rolled into 1182.17.
- Total: Total of all reporting groups
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients) | Total
Number analyzed (Participants) | 291 | 255 | 449 | 995
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (8) | 45.6 (8.2) | 43.5 (7.7) | 44.1 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 20 | 44 | 99
  Male | 256 | 235 | 405 | 896

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Haemoglobin
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: FAS17 - Group 1: TPV/r patients who rolled over from Trials 1182.2, 1182.4, 1182.6, 1182.52, 1182.12 and 1182.48 Group 2: Patients from 1182.51 who rolled over into 1182.17 Group 3: PI comparator arm patients from 1182.4, 1182.12 and 1182.48 who virologically failed and who then rolled into 1182.17.
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 1 [-2.41 to -0.30] | 2 [-1.56 to -0.17] | 6 [-1.37 to -0.07]

2. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - White Blood Cell ct.
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 5 | 14 | 20

3. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Platelets
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 9 | 7 | 7

4. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Prothrombin Time
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 4 | 0 | 0

5. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Sodium
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 2 | 0 | 1

6. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Potassium
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 5 | 1 | 3

7. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Calcium
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 6 | 1 | 2

8. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Phosphate
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 8 | 0 | 0

9. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Carbon Dioxide
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 4 | 0 | 2

10. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Aspartate Aminotransferase (AST/GOT,SGOT)
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 24 | 13 | 22

11. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Alanine Aminotransferase (ALT/GPT,SGPT)
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 47 | 27 | 42

12. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Alkaline Phosphatase
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 1 | 0 | 2

13. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Amylase
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 31 | 24 | 48

14. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Creatine Phosphokinase
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 14 | 8 | 17

15. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Lipase
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 16 | 8 | 12

16. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Glucose
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 10 | 2 | 7

17. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Cholesterol, Total
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 82 | 34 | 30

18. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Creatinine
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 5 | 6 | 10

19. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Bilirubin, Total
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 4 | 1 | 1

20. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Triglycerides
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 75 | 57 | 38

21. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Uric Acid
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 2 | 0 | 5

22. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 - Albumin
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 0 | 0 | 0

23. Primary Outcome: Number of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 -Low-density Lipoprotein (LDL)
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 48 | 15 | 12

24. Primary Outcome: Number of Patients With Adverse Events Leading to Death
Description: NIH Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: End of Trial (>288 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
participants | 10 | 13 | 26

25. Secondary Outcome: Change From Baseline in Human Immunodeficiency Virus-Ribonucleic Acid (HIV-RNA) Viral Load - Last Observation Carried Forward (LOCF)
Description: Change from baseline in Human Immunodeficiency Virus-Ribonucleic Acid (HIV-RNA) viral load with last observation carried forward (LOCF)
Time Frame: Baseline to 192-240 week time interval
Population: FAS17 with last observation carried forward (LOCF, missing were replaced by the previous non-missing value), Group 1: TPV/r patients from Trials 1182.2, 1182.4, 1182.6, 1182.52, 1182.12 and 1182.48; Group 2: Patients from 1182.51; Group 3: PI comparator arm patients from 1182.4, 1182.12 and 1182.48 who virologically failed and rolled into 1182.17
Measure: Median (Inter-Quartile Range); unit: Log 10 copies/mL
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 291 | 255 | 449
Log 10 copies/mL | -1.19 [-2.41 to 0.30] | -0.62 [-1.56 to -0.17] | -0.5 [-1.37 to -0.07]

26. Secondary Outcome: Change From Baseline in CD4 Cell Count (LOCF)
Description: Change from baseline in CD4 cell count with last observation carried forward(LOCF).
Time Frame: Baseline to 192-240 week time interval
Population: FAS17 with last observation carried forward (LOCF, missing were replaced by the previous non-missing value), Group 1: TPV/r patients from Trials 1182.2, 1182.4,1182.6, 1182.52, 1182.12 and 1182.48; Group 2: Patients from 1182.51; Group 3: PI comparator arm patients from 1182.4, 1182.12 and 1182.48 who virologically failed.
Measure: Mean (Standard Deviation); unit: cells/mm3
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Number analyzed (Participants) | 240 | 253 | 449
cells/mm3 | 83 (178) | 26 (149) | 21 (132)

ADVERSE EVENTS:
Time Frame: Up to 288 weeks. From the time patients received their first dose of TPV/r until the last patient out of the study on 26 May 2008 (for those patients who entered Trial 1182.17).
Arm/Group | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Serious Adverse Events (participants affected / at risk) | 100 | 91 | 135
Other Adverse Events (participants affected / at risk) | 284 | 250 | 406
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Anaemia (Blood and lymphatic system disorders) | 5/291 | 10/255 | 9/449
Eosinophilia (Blood and lymphatic system disorders) | 0/291 | 0/255 | 1/449
Febrile neutropenia (Blood and lymphatic system disorders) | 1/291 | 2/255 | 1/449
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0/291 | 0/255 | 1/449
Leukopenia (Blood and lymphatic system disorders) | 1/291 | 0/255 | 0/449
Lymphadenopathy (Blood and lymphatic system disorders) | 0/291 | 1/255 | 0/449
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 0/291 | 1/255 | 0/449
Neutropenia (Blood and lymphatic system disorders) | 2/291 | 0/255 | 1/449
Pancytopenia (Blood and lymphatic system disorders) | 0/291 | 1/255 | 2/449
Thrombocytopenia (Blood and lymphatic system disorders) | 1/291 | 0/255 | 0/449
Acute myocardial infarction (Cardiac disorders) | 1/291 | 1/255 | 0/449
Angina pectoris (Cardiac disorders) | 1/291 | 1/255 | 0/449
Angina unstable (Cardiac disorders) | 2/291 | 2/255 | 0/449
Arrhythmia (Cardiac disorders) | 0/291 | 0/255 | 1/449
Atrial fibrillation (Cardiac disorders) | 1/291 | 1/255 | 0/449
Cardiac arrest (Cardiac disorders) | 0/291 | 0/255 | 1/449
Cardiac failure (Cardiac disorders) | 0/291 | 1/255 | 1/449
Cardiac failure congestive (Cardiac disorders) | 1/291 | 1/255 | 1/449
Cardiac tamponade (Cardiac disorders) | 1/291 | 0/255 | 0/449
Cardio-respiratory arrest (Cardiac disorders) | 1/291 | 1/255 | 2/449
Cardiopulmonary failure (Cardiac disorders) | 0/291 | 0/255 | 1/449
Cor pulmonale (Cardiac disorders) | 1/291 | 0/255 | 0/449
Coronary artery disease (Cardiac disorders) | 1/291 | 1/255 | 0/449
Intracardiac thrombus (Cardiac disorders) | 1/291 | 0/255 | 0/449
Ischaemic cardiomyopathy (Cardiac disorders) | 0/291 | 2/255 | 0/449
Myocardial infarction (Cardiac disorders) | 2/291 | 2/255 | 0/449
Right ventricular failure (Cardiac disorders) | 0/291 | 0/255 | 1/449
Tachycardia (Cardiac disorders) | 1/291 | 1/255 | 1/449
Ventricular tachycardia (Cardiac disorders) | 0/291 | 0/255 | 1/449
Fanconi syndrome (Congenital, familial and genetic disorders) | 1/291 | 0/255 | 0/449
Ear pain (Ear and labyrinth disorders) | 1/291 | 0/255 | 0/449
Cataract (Eye disorders) | 0/291 | 2/255 | 0/449
Retinal artery embolism (Eye disorders) | 0/291 | 1/255 | 0/449
Retinal detachment (Eye disorders) | 1/291 | 0/255 | 1/449
Vision blurred (Eye disorders) | 0/291 | 1/255 | 0/449
Abdominal hernia (Gastrointestinal disorders) | 0/291 | 0/255 | 1/449
Abdominal pain (Gastrointestinal disorders) | 5/291 | 2/255 | 8/449
Abdominal pain upper (Gastrointestinal disorders) | 1/291 | 0/255 | 1/449
Anal haemorrhage (Gastrointestinal disorders) | 0/291 | 0/255 | 1/449
Anal ulcer (Gastrointestinal disorders) | 1/291 | 0/255 | 1/449
Aphthous stomatitis (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Appendicitis perforated (Gastrointestinal disorders) | 0/291 | 1/255 | 0/449
Constipation (Gastrointestinal disorders) | 1/291 | 1/255 | 0/449
Diarrhoea (Gastrointestinal disorders) | 10/291 | 5/255 | 7/449
Diverticular perforation (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Diverticulum (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Enteritis (Gastrointestinal disorders) | 0/291 | 1/255 | 0/449
Faecal incontinence (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Faeces discoloured (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Gastritis (Gastrointestinal disorders) | 0/291 | 1/255 | 1/449
Gastrointestinal disorder (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2/291 | 2/255 | 0/449
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Haemorrhoids (Gastrointestinal disorders) | 0/291 | 0/255 | 2/449
Impaired gastric emptying (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Inguinal hernia (Gastrointestinal disorders) | 1/291 | 1/255 | 0/449
Intestinal perforation (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Irritable bowel syndrome (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Lip ulceration (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Nausea (Gastrointestinal disorders) | 2/291 | 3/255 | 3/449
Oesophageal pain (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Oesophageal stenosis (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Oesophageal ulcer (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Oesophagitis (Gastrointestinal disorders) | 1/291 | 0/255 | 1/449
Oral disorder (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Oral pain (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Pancreatitis (Gastrointestinal disorders) | 1/291 | 2/255 | 3/449
Pancreatitis acute (Gastrointestinal disorders) | 0/291 | 2/255 | 2/449
Peptic ulcer (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Peritoneal adhesions (Gastrointestinal disorders) | 1/291 | 0/255 | 0/449
Proctitis (Gastrointestinal disorders) | 0/291 | 0/255 | 1/449
Rectal haemorrhage (Gastrointestinal disorders) | 2/291 | 0/255 | 1/449
Vomiting (Gastrointestinal disorders) | 3/291 | 4/255 | 4/449
Adverse drug reaction (General disorders) | 0/291 | 1/255 | 0/449
Asthenia (General disorders) | 1/291 | 2/255 | 6/449
Chest pain (General disorders) | 6/291 | 3/255 | 3/449
Chills (General disorders) | 0/291 | 1/255 | 1/449
Cyst (General disorders) | 1/291 | 0/255 | 0/449
Death (General disorders) | 0/291 | 1/255 | 0/449
Drug withdrawal syndrome (General disorders) | 0/291 | 1/255 | 0/449
Fatigue (General disorders) | 0/291 | 1/255 | 2/449
General physical health deterioration (General disorders) | 1/291 | 2/255 | 2/449
Generalised oedema (General disorders) | 1/291 | 0/255 | 1/449
Influenza like illness (General disorders) | 0/291 | 0/255 | 1/449
Local swelling (General disorders) | 1/291 | 0/255 | 0/449
Malaise (General disorders) | 2/291 | 0/255 | 2/449
Multi-organ failure (General disorders) | 0/291 | 2/255 | 3/449
Oedema peripheral (General disorders) | 1/291 | 1/255 | 0/449
Pain (General disorders) | 2/291 | 0/255 | 1/449
Polyserositis (General disorders) | 0/291 | 1/255 | 0/449
Pyrexia (General disorders) | 14/291 | 13/255 | 19/449
Acute hepatic failure (Hepatobiliary disorders) | 0/291 | 0/255 | 1/449
Cholangitis (Hepatobiliary disorders) | 0/291 | 0/255 | 1/449
Cholecystitis (Hepatobiliary disorders) | 1/291 | 3/255 | 1/449
Cholelithiasis (Hepatobiliary disorders) | 1/291 | 1/255 | 0/449
Cytolytic hepatitis (Hepatobiliary disorders) | 0/291 | 1/255 | 1/449
Hepatic failure (Hepatobiliary disorders) | 0/291 | 0/255 | 1/449
Hepatosplenomegaly (Hepatobiliary disorders) | 0/291 | 0/255 | 1/449
Hepatotoxicity (Hepatobiliary disorders) | 0/291 | 0/255 | 1/449
Hyperbilirubinaemia (Hepatobiliary disorders) | 1/291 | 0/255 | 0/449
Jaundice (Hepatobiliary disorders) | 0/291 | 2/255 | 0/449
Jaundice cholestatic (Hepatobiliary disorders) | 1/291 | 0/255 | 0/449
Liver injury (Hepatobiliary disorders) | 0/291 | 0/255 | 1/449
Anaphylactic shock (Immune system disorders) | 1/291 | 0/255 | 0/449
Drug hypersensitivity (Immune system disorders) | 0/291 | 0/255 | 2/449
Immune reconstitution syndrome (Immune system disorders) | 0/291 | 0/255 | 1/449
Immunodeficiency (Immune system disorders) | 0/291 | 0/255 | 1/449
AIDS dementia complex (Infections and infestations) | 0/291 | 0/255 | 1/449
AIDS encephalopathy (Infections and infestations) | 0/291 | 0/255 | 1/449
Abdominal wall abscess (Infections and infestations) | 0/291 | 0/255 | 1/449
Abscess (Infections and infestations) | 0/291 | 0/255 | 2/449
Abscess limb (Infections and infestations) | 1/291 | 0/255 | 0/449
Abscess neck (Infections and infestations) | 1/291 | 0/255 | 0/449
Acanthamoeba infection (Infections and infestations) | 1/291 | 0/255 | 0/449
Acquired immunodeficiency syndrome (Infections and infestations) | 0/291 | 1/255 | 1/449
Anal abscess (Infections and infestations) | 1/291 | 2/255 | 1/449
Anogenital warts (Infections and infestations) | 2/291 | 0/255 | 1/449
Anorectal cellulitis (Infections and infestations) | 1/291 | 0/255 | 0/449
Appendiceal abscess (Infections and infestations) | 1/291 | 0/255 | 0/449
Appendicitis (Infections and infestations) | 0/291 | 0/255 | 4/449
Arthritis bacterial (Infections and infestations) | 0/291 | 0/255 | 1/449
Aspergillosis (Infections and infestations) | 0/291 | 1/255 | 0/449
Bacteraemia (Infections and infestations) | 1/291 | 0/255 | 1/449
Bacterial sepsis (Infections and infestations) | 1/291 | 0/255 | 0/449
Bronchitis (Infections and infestations) | 2/291 | 3/255 | 0/449
Campylobacter intestinal infection (Infections and infestations) | 0/291 | 1/255 | 2/449
Catheter related infection (Infections and infestations) | 1/291 | 0/255 | 3/449
Cellulitis (Infections and infestations) | 3/291 | 1/255 | 2/449
Cellulitis of male external genital organ (Infections and infestations) | 1/291 | 0/255 | 0/449
Central line infection (Infections and infestations) | 1/291 | 1/255 | 0/449
Cerebral toxoplasmosis (Infections and infestations) | 1/291 | 0/255 | 2/449
Choriomeningitis lymphocytic (Infections and infestations) | 1/291 | 0/255 | 0/449
Chronic sinusitis (Infections and infestations) | 0/291 | 0/255 | 1/449
Clostridial infection (Infections and infestations) | 0/291 | 0/255 | 1/449
Cryptosporidiosis infection (Infections and infestations) | 0/291 | 0/255 | 1/449
Cytomegalovirus chorioretinitis (Infections and infestations) | 1/291 | 1/255 | 2/449
Cytomegalovirus colitis (Infections and infestations) | 1/291 | 0/255 | 0/449
Cytomegalovirus infection (Infections and infestations) | 2/291 | 1/255 | 0/449
Cytomegalovirus oesophagitis (Infections and infestations) | 0/291 | 0/255 | 1/449
Cytomegalovirus viraemia (Infections and infestations) | 0/291 | 0/255 | 1/449
Diarrhoea infectious (Infections and infestations) | 1/291 | 0/255 | 0/449
Encephalitis cytomegalovirus (Infections and infestations) | 1/291 | 0/255 | 1/449
Encephalitis herpes (Infections and infestations) | 0/291 | 0/255 | 1/449
Encephalitis viral (Infections and infestations) | 0/291 | 0/255 | 1/449
End stage AIDS (Infections and infestations) | 0/291 | 0/255 | 1/449
Endocarditis bacterial (Infections and infestations) | 0/291 | 0/255 | 1/449
Enterocolitis infectious (Infections and infestations) | 0/291 | 0/255 | 1/449
Escherichia urinary tract infection (Infections and infestations) | 1/291 | 0/255 | 0/449
Fungal oesophagitis (Infections and infestations) | 0/291 | 0/255 | 2/449
Gastritis fungal (Infections and infestations) | 0/291 | 0/255 | 1/449
Gastroenteritis (Infections and infestations) | 0/291 | 0/255 | 1/449
Giardiasis (Infections and infestations) | 1/291 | 0/255 | 0/449
Groin abscess (Infections and infestations) | 0/291 | 0/255 | 1/449
HIV infection (Infections and infestations) | 0/291 | 3/255 | 1/449
Hepatitis viral (Infections and infestations) | 0/291 | 0/255 | 1/449
Herpes oesophagitis (Infections and infestations) | 0/291 | 0/255 | 1/449
Herpes simplex (Infections and infestations) | 0/291 | 0/255 | 1/449
Herpes zoster (Infections and infestations) | 0/291 | 1/255 | 0/449
Infection (Infections and infestations) | 1/291 | 0/255 | 1/449
Klebsiella bacteraemia (Infections and infestations) | 0/291 | 1/255 | 0/449
Klebsiella sepsis (Infections and infestations) | 0/291 | 1/255 | 0/449
Lobar pneumonia (Infections and infestations) | 2/291 | 3/255 | 1/449
Lower respiratory tract infection (Infections and infestations) | 1/291 | 1/255 | 0/449
Lung abscess (Infections and infestations) | 0/291 | 0/255 | 1/449
Lymph node tuberculosis (Infections and infestations) | 0/291 | 0/255 | 1/449
Mediastinitis (Infections and infestations) | 0/291 | 0/255 | 1/449
Meningitis cryptococcal (Infections and infestations) | 1/291 | 0/255 | 1/449
Meningitis pneumococcal (Infections and infestations) | 0/291 | 0/255 | 1/449
Molluscum contagiosum (Infections and infestations) | 0/291 | 0/255 | 1/449
Mycobacterial infection (Infections and infestations) | 1/291 | 0/255 | 1/449
Mycobacterium avium complex infection (Infections and infestations) | 3/291 | 0/255 | 3/449
Necrotising herpetic retinopathy (Infections and infestations) | 0/291 | 1/255 | 0/449
Oesophageal candidiasis (Infections and infestations) | 3/291 | 2/255 | 4/449
Oral candidiasis (Infections and infestations) | 1/291 | 1/255 | 3/449
Orchitis (Infections and infestations) | 1/291 | 1/255 | 0/449
Papilloma viral infection (Infections and infestations) | 0/291 | 0/255 | 1/449
Perineal abscess (Infections and infestations) | 1/291 | 0/255 | 0/449
Perirectal abscess (Infections and infestations) | 0/291 | 2/255 | 0/449
Pneumococcal infection (Infections and infestations) | 0/291 | 1/255 | 0/449
Pneumococcal sepsis (Infections and infestations) | 1/291 | 0/255 | 0/449
Pneumocystis jiroveci pneumonia (Infections and infestations) | 2/291 | 1/255 | 8/449
Pneumonia (Infections and infestations) | 6/291 | 9/255 | 9/449
Pneumonia bacterial (Infections and infestations) | 1/291 | 2/255 | 1/449
Pneumonia cytomegaloviral (Infections and infestations) | 1/291 | 1/255 | 0/449
Pneumonia necrotising (Infections and infestations) | 0/291 | 0/255 | 1/449
Pneumonia pneumococcal (Infections and infestations) | 0/291 | 0/255 | 2/449
Pneumonia staphylococcal (Infections and infestations) | 0/291 | 1/255 | 1/449
Postoperative wound infection (Infections and infestations) | 1/291 | 0/255 | 0/449
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0/291 | 4/255 | 1/449
Pseudomembranous colitis (Infections and infestations) | 1/291 | 0/255 | 0/449
Pseudomonal sepsis (Infections and infestations) | 0/291 | 1/255 | 0/449
Pulmonary tuberculosis (Infections and infestations) | 0/291 | 0/255 | 1/449
Pyelonephritis (Infections and infestations) | 0/291 | 1/255 | 0/449
Rectal abscess (Infections and infestations) | 1/291 | 2/255 | 0/449
Respiratory tract infection viral (Infections and infestations) | 0/291 | 0/255 | 1/449
Scrotal abscess (Infections and infestations) | 1/291 | 0/255 | 0/449
Sepsis (Infections and infestations) | 3/291 | 1/255 | 2/449
Septic shock (Infections and infestations) | 1/291 | 0/255 | 2/449
Sinusitis (Infections and infestations) | 4/291 | 0/255 | 1/449
Sinusitis aspergillus (Infections and infestations) | 0/291 | 1/255 | 0/449
Sinusitis bacterial (Infections and infestations) | 0/291 | 1/255 | 0/449
Staphylococcal infection (Infections and infestations) | 3/291 | 2/255 | 1/449
Staphylococcal sepsis (Infections and infestations) | 1/291 | 0/255 | 0/449
Streptococcal infection (Infections and infestations) | 0/291 | 0/255 | 1/449
Streptococcal sepsis (Infections and infestations) | 0/291 | 0/255 | 1/449
Subcutaneous abscess (Infections and infestations) | 1/291 | 0/255 | 0/449
Syphilis (Infections and infestations) | 0/291 | 0/255 | 1/449
Urinary tract infection (Infections and infestations) | 1/291 | 0/255 | 0/449
Urinary tract infection enterococcal (Infections and infestations) | 0/291 | 1/255 | 0/449
Viral infection (Infections and infestations) | 0/291 | 0/255 | 2/449
Viral sinusitis (Infections and infestations) | 1/291 | 0/255 | 0/449
Viral upper respiratory tract infection (Infections and infestations) | 0/291 | 1/255 | 0/449
Burns third degree (Injury, poisoning and procedural complications) | 1/291 | 0/255 | 0/449
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 1/291 | 0/255 | 0/449
Fall (Injury, poisoning and procedural complications) | 1/291 | 0/255 | 1/449
Femur fracture (Injury, poisoning and procedural complications) | 1/291 | 0/255 | 0/449
Head injury (Injury, poisoning and procedural complications) | 1/291 | 0/255 | 0/449
Hip fracture (Injury, poisoning and procedural complications) | 1/291 | 0/255 | 0/449
Injury (Injury, poisoning and procedural complications) | 0/291 | 0/255 | 1/449
Joint dislocation (Injury, poisoning and procedural complications) | 1/291 | 0/255 | 0/449
Lower limb fracture (Injury, poisoning and procedural complications) | 0/291 | 0/255 | 1/449
Neck injury (Injury, poisoning and procedural complications) | 1/291 | 0/255 | 0/449
Overdose (Injury, poisoning and procedural complications) | 1/291 | 0/255 | 0/449
Patella fracture (Injury, poisoning and procedural complications) | 1/291 | 1/255 | 0/449
Post procedural haematoma (Injury, poisoning and procedural complications) | 1/291 | 0/255 | 0/449
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1/291 | 0/255 | 1/449
Road traffic accident (Injury, poisoning and procedural complications) | 1/291 | 2/255 | 2/449
Skeletal injury (Injury, poisoning and procedural complications) | 0/291 | 1/255 | 0/449
Spinal compression fracture (Injury, poisoning and procedural complications) | 0/291 | 1/255 | 0/449
Splenic rupture (Injury, poisoning and procedural complications) | 0/291 | 1/255 | 0/449
Stress fracture (Injury, poisoning and procedural complications) | 1/291 | 0/255 | 0/449
Tendon rupture (Injury, poisoning and procedural complications) | 1/291 | 0/255 | 0/449
Transfusion reaction (Injury, poisoning and procedural complications) | 0/291 | 1/255 | 0/449
Traumatic brain injury (Injury, poisoning and procedural complications) | 0/291 | 0/255 | 1/449
Upper limb fracture (Injury, poisoning and procedural complications) | 0/291 | 1/255 | 0/449
Wound (Injury, poisoning and procedural complications) | 0/291 | 1/255 | 0/449
Alanine aminotransferase increased (Investigations) | 0/291 | 0/255 | 2/449
Aspartate aminotransferase increased (Investigations) | 0/291 | 0/255 | 2/449
Biopsy breast (Investigations) | 0/291 | 0/255 | 1/449
Blood bilirubin increased (Investigations) | 0/291 | 1/255 | 1/449
Blood creatine phosphokinase increased (Investigations) | 0/291 | 1/255 | 0/449
Blood creatinine increased (Investigations) | 1/291 | 1/255 | 0/449
Blood lactate dehydrogenase increased (Investigations) | 0/291 | 0/255 | 1/449
Blood urea increased (Investigations) | 1/291 | 0/255 | 0/449
Fungus serology test positive (Investigations) | 1/291 | 0/255 | 0/449
Gamma-glutamyltransferase increased (Investigations) | 1/291 | 1/255 | 1/449
Haematocrit decreased (Investigations) | 0/291 | 0/255 | 1/449
Haemoglobin decreased (Investigations) | 0/291 | 0/255 | 1/449
Hepatic enzyme increased (Investigations) | 0/291 | 3/255 | 0/449
Liver function test abnormal (Investigations) | 1/291 | 1/255 | 1/449
Liver scan abnormal (Investigations) | 0/291 | 0/255 | 1/449
Transaminases increased (Investigations) | 0/291 | 1/255 | 0/449
Weight decreased (Investigations) | 1/291 | 0/255 | 2/449
Cachexia (Metabolism and nutrition disorders) | 1/291 | 2/255 | 5/449
Dehydration (Metabolism and nutrition disorders) | 4/291 | 4/255 | 9/449
Electrolyte imbalance (Metabolism and nutrition disorders) | 1/291 | 0/255 | 0/449
Failure to thrive (Metabolism and nutrition disorders) | 0/291 | 0/255 | 1/449
Fat redistribution (Metabolism and nutrition disorders) | 1/291 | 0/255 | 0/449
Malnutrition (Metabolism and nutrition disorders) | 0/291 | 0/255 | 1/449
Metabolic acidosis (Metabolism and nutrition disorders) | 0/291 | 1/255 | 2/449
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/291 | 1/255 | 0/449
Arthropathy (Musculoskeletal and connective tissue disorders) | 0/291 | 0/255 | 1/449
Back pain (Musculoskeletal and connective tissue disorders) | 1/291 | 0/255 | 2/449
Bone erosion (Musculoskeletal and connective tissue disorders) | 0/291 | 1/255 | 0/449
Flank pain (Musculoskeletal and connective tissue disorders) | 1/291 | 0/255 | 0/449
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1/291 | 0/255 | 0/449
Neck pain (Musculoskeletal and connective tissue disorders) | 1/291 | 0/255 | 0/449
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/291 | 0/255 | 1/449
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 6/291 | 0/255 | 0/449
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0/291 | 0/255 | 1/449
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/291 | 0/255 | 0/449
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1/291 | 0/255 | 0/449
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0/291 | 1/255 | 0/449
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/291 | 0/255 | 0/449
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1/291 | 0/255 | 0/449
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/291 | 1/255 | 0/449
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/291 | 1/255 | 2/449
Anal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/291 | 0/255 | 1/449
Anal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/291 | 1/255 | 1/449
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/291 | 0/255 | 0/449
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/291 | 1/255 | 2/449
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/291 | 0/255 | 1/449
Bowenoid papulosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/291 | 1/255 | 0/449
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/291 | 1/255 | 1/449
Colorectal carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/291 | 0/255 | 0/449
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/291 | 0/255 | 1/449
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/291 | 1/255 | 1/449
Hodgkin's disease stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/291 | 0/255 | 0/449
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/291 | 1/255 | 3/449
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/291 | 1/255 | 0/449
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/291 | 0/255 | 1/449
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/291 | 1/255 | 1/449
Malignant anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/291 | 0/255 | 1/449
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/291 | 0/255 | 1/449
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/291 | 1/255 | 0/449
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/291 | 0/255 | 1/449
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/291 | 1/255 | 0/449
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/291 | 0/255 | 1/449
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/291 | 0/255 | 0/449
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/291 | 0/255 | 1/449
Splenic neoplasm malignancy unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/291 | 0/255 | 0/449
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/291 | 0/255 | 0/449
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/291 | 0/255 | 1/449
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/291 | 0/255 | 0/449
Brain oedema (Nervous system disorders) | 0/291 | 0/255 | 1/449
Carotid artery stenosis (Nervous system disorders) | 0/291 | 1/255 | 0/449
Carpal tunnel syndrome (Nervous system disorders) | 0/291 | 1/255 | 0/449
Cerebral haematoma (Nervous system disorders) | 0/291 | 0/255 | 1/449
Cerebral haemorrhage (Nervous system disorders) | 1/291 | 0/255 | 0/449
Cerebrovascular accident (Nervous system disorders) | 1/291 | 0/255 | 0/449
Convulsion (Nervous system disorders) | 1/291 | 1/255 | 3/449
Encephalitis (Nervous system disorders) | 0/291 | 1/255 | 0/449
Epilepsy (Nervous system disorders) | 0/291 | 1/255 | 0/449
Facial palsy (Nervous system disorders) | 1/291 | 0/255 | 0/449
Haemorrhage intracranial (Nervous system disorders) | 1/291 | 0/255 | 1/449
Headache (Nervous system disorders) | 1/291 | 1/255 | 5/449
Hypertensive encephalopathy (Nervous system disorders) | 1/291 | 0/255 | 0/449
Intracranial aneurysm (Nervous system disorders) | 1/291 | 0/255 | 0/449
Intracranial hypotension (Nervous system disorders) | 0/291 | 1/255 | 0/449
Ischaemic stroke (Nervous system disorders) | 1/291 | 0/255 | 0/449
Lethargy (Nervous system disorders) | 0/291 | 0/255 | 1/449
Leukoencephalopathy (Nervous system disorders) | 1/291 | 0/255 | 0/449
Loss of consciousness (Nervous system disorders) | 0/291 | 0/255 | 1/449
Memory impairment (Nervous system disorders) | 0/291 | 1/255 | 0/449
Nervous system disorder (Nervous system disorders) | 0/291 | 0/255 | 1/449
Neuropathy peripheral (Nervous system disorders) | 0/291 | 1/255 | 0/449
Paraesthesia (Nervous system disorders) | 0/291 | 0/255 | 1/449
Sinus headache (Nervous system disorders) | 0/291 | 1/255 | 0/449
Syncope (Nervous system disorders) | 3/291 | 0/255 | 0/449
Transient ischaemic attack (Nervous system disorders) | 0/291 | 0/255 | 1/449
Tremor (Nervous system disorders) | 1/291 | 0/255 | 0/449
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/291 | 0/255 | 1/449
Anxiety disorder (Psychiatric disorders) | 0/291 | 1/255 | 0/449
Completed suicide (Psychiatric disorders) | 1/291 | 0/255 | 0/449
Confusional state (Psychiatric disorders) | 1/291 | 1/255 | 1/449
Depression (Psychiatric disorders) | 3/291 | 2/255 | 1/449
Drug abuse (Psychiatric disorders) | 2/291 | 0/255 | 0/449
Hallucination (Psychiatric disorders) | 0/291 | 0/255 | 1/449
Hallucination, tactile (Psychiatric disorders) | 1/291 | 0/255 | 0/449
Hypomania (Psychiatric disorders) | 1/291 | 0/255 | 0/449
Mental status changes (Psychiatric disorders) | 0/291 | 0/255 | 1/449
Paranoia (Psychiatric disorders) | 1/291 | 0/255 | 0/449
Suicide attempt (Psychiatric disorders) | 2/291 | 0/255 | 1/449
Withdrawal syndrome (Psychiatric disorders) | 0/291 | 1/255 | 0/449
Calculus ureteric (Renal and urinary disorders) | 0/291 | 0/255 | 1/449
Focal glomerulosclerosis (Renal and urinary disorders) | 0/291 | 0/255 | 1/449
Glomerulonephritis proliferative (Renal and urinary disorders) | 0/291 | 0/255 | 1/449
Nephritis interstitial (Renal and urinary disorders) | 0/291 | 1/255 | 0/449
Nephrolithiasis (Renal and urinary disorders) | 1/291 | 0/255 | 0/449
Oliguria (Renal and urinary disorders) | 0/291 | 0/255 | 1/449
Renal colic (Renal and urinary disorders) | 1/291 | 0/255 | 0/449
Renal failure (Renal and urinary disorders) | 3/291 | 3/255 | 4/449
Renal failure acute (Renal and urinary disorders) | 8/291 | 2/255 | 4/449
Renal impairment (Renal and urinary disorders) | 0/291 | 0/255 | 2/449
Renal tubular acidosis (Renal and urinary disorders) | 1/291 | 0/255 | 0/449
Renal tubular disorder (Renal and urinary disorders) | 0/291 | 1/255 | 1/449
Renal tubular necrosis (Renal and urinary disorders) | 0/291 | 0/255 | 1/449
Breast pain (Reproductive system and breast disorders) | 0/291 | 0/255 | 1/449
Cervical dysplasia (Reproductive system and breast disorders) | 0/291 | 0/255 | 1/449
Epididymitis (Reproductive system and breast disorders) | 0/291 | 0/255 | 1/449
Fallopian tube obstruction (Reproductive system and breast disorders) | 0/291 | 0/255 | 1/449
Haematosalpinx (Reproductive system and breast disorders) | 0/291 | 0/255 | 1/449
Metrorrhagia (Reproductive system and breast disorders) | 0/291 | 0/255 | 1/449
Prostatitis (Reproductive system and breast disorders) | 1/291 | 1/255 | 1/449
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0/291 | 1/255 | 0/449
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/291 | 0/255 | 0/449
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0/291 | 0/255 | 1/449
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/291 | 2/255 | 1/449
Cough (Respiratory, thoracic and mediastinal disorders) | 0/291 | 0/255 | 2/449
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/291 | 4/255 | 2/449
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0/291 | 0/255 | 1/449
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0/291 | 1/255 | 2/449
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0/291 | 0/255 | 1/449
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0/291 | 1/255 | 0/449
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0/291 | 2/255 | 3/449
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0/291 | 0/255 | 1/449
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0/291 | 0/255 | 1/449
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0/291 | 0/255 | 1/449
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0/291 | 0/255 | 1/449
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/291 | 1/255 | 0/449
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1/291 | 0/255 | 0/449
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0/291 | 0/255 | 1/449
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0/291 | 0/255 | 1/449
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/291 | 2/255 | 1/449
Snoring (Respiratory, thoracic and mediastinal disorders) | 0/291 | 0/255 | 1/449
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0/291 | 0/255 | 1/449
Drug eruption (Skin and subcutaneous tissue disorders) | 0/291 | 1/255 | 1/449
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 1/291 | 2/255 | 0/449
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 2/291 | 1/255 | 0/449
Rash (Skin and subcutaneous tissue disorders) | 1/291 | 0/255 | 0/449
Rash pruritic (Skin and subcutaneous tissue disorders) | 0/291 | 2/255 | 0/449
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0/291 | 0/255 | 1/449
Skin lesion (Skin and subcutaneous tissue disorders) | 1/291 | 0/255 | 0/449
Skin toxicity (Skin and subcutaneous tissue disorders) | 0/291 | 0/255 | 1/449
Colostomy (Surgical and medical procedures) | 1/291 | 0/255 | 0/449
Intestinal anastomosis (Surgical and medical procedures) | 1/291 | 0/255 | 0/449
Intestinal operation (Surgical and medical procedures) | 1/291 | 0/255 | 0/449
Lymphadenectomy (Surgical and medical procedures) | 0/291 | 0/255 | 1/449
Umbilical hernia repair (Surgical and medical procedures) | 1/291 | 0/255 | 0/449
Wisdom teeth removal (Surgical and medical procedures) | 0/291 | 0/255 | 1/449
Air embolism (Vascular disorders) | 0/291 | 0/255 | 1/449
Arteriosclerosis (Vascular disorders) | 1/291 | 0/255 | 0/449
Deep vein thrombosis (Vascular disorders) | 0/291 | 0/255 | 1/449
Hypertension (Vascular disorders) | 0/291 | 1/255 | 3/449
Hypotension (Vascular disorders) | 1/291 | 0/255 | 2/449
Hypovolaemic shock (Vascular disorders) | 1/291 | 0/255 | 0/449
Lymphocele (Vascular disorders) | 0/291 | 1/255 | 0/449
Necrosis ischaemic (Vascular disorders) | 1/291 | 0/255 | 0/449
Varicose vein (Vascular disorders) | 0/291 | 0/255 | 1/449
Venous occlusion (Vascular disorders) | 1/291 | 0/255 | 0/449
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Group 1 (Patients With Varying Degrees of Treatment Experience | Group 2 (Highly Treatment Experienced Patients) | Group 3 (Tipranavir naïve Patients)
Anaemia (Blood and lymphatic system disorders) | 22/291 | 22/255 | 19/449
Lymphadenopathy (Blood and lymphatic system disorders) | 18/291 | 11/255 | 20/449
Abdominal distension (Gastrointestinal disorders) | 15/291 | 5/255 | 9/449
Abdominal pain (Gastrointestinal disorders) | 45/291 | 26/255 | 42/449
Abdominal pain upper (Gastrointestinal disorders) | 17/291 | 18/255 | 16/449
Constipation (Gastrointestinal disorders) | 21/291 | 13/255 | 13/449
Diarrhoea (Gastrointestinal disorders) | 152/291 | 107/255 | 126/449
Dyspepsia (Gastrointestinal disorders) | 21/291 | 16/255 | 9/449
Flatulence (Gastrointestinal disorders) | 19/291 | 18/255 | 23/449
Haemorrhoids (Gastrointestinal disorders) | 15/291 | 6/255 | 15/449
Nausea (Gastrointestinal disorders) | 101/291 | 62/255 | 72/449
Vomiting (Gastrointestinal disorders) | 56/291 | 30/255 | 35/449
Adverse drug reaction (General disorders) | 9/291 | 27/255 | 34/449
Asthenia (General disorders) | 27/291 | 28/255 | 35/449
Chest pain (General disorders) | 18/291 | 9/255 | 11/449
Fatigue (General disorders) | 80/291 | 58/255 | 47/449
Influenza like illness (General disorders) | 17/291 | 11/255 | 10/449
Injection site reaction (General disorders) | 12/291 | 22/255 | 24/449
Pain (General disorders) | 18/291 | 5/255 | 9/449
Pyrexia (General disorders) | 53/291 | 44/255 | 59/449
Anogenital warts (Infections and infestations) | 17/291 | 12/255 | 9/449
Bronchitis (Infections and infestations) | 42/291 | 39/255 | 42/449
Folliculitis (Infections and infestations) | 18/291 | 8/255 | 9/449
Gastroenteritis (Infections and infestations) | 12/291 | 18/255 | 17/449
Herpes simplex (Infections and infestations) | 15/291 | 8/255 | 14/449
Herpes zoster (Infections and infestations) | 23/291 | 10/255 | 20/449
Influenza (Infections and infestations) | 31/291 | 18/255 | 29/449
Nasopharyngitis (Infections and infestations) | 54/291 | 43/255 | 60/449
Oesophageal candidiasis (Infections and infestations) | 7/291 | 17/255 | 17/449
Onychomycosis (Infections and infestations) | 19/291 | 9/255 | 13/449
Oral candidiasis (Infections and infestations) | 27/291 | 34/255 | 43/449
Oral herpes (Infections and infestations) | 17/291 | 14/255 | 18/449
Rhinitis (Infections and infestations) | 20/291 | 14/255 | 10/449
Sinusitis (Infections and infestations) | 48/291 | 29/255 | 33/449
Upper respiratory tract infection (Infections and infestations) | 76/291 | 27/255 | 36/449
Urinary tract infection (Infections and infestations) | 23/291 | 8/255 | 15/449
Weight decreased (Investigations) | 27/291 | 20/255 | 26/449
Anorexia (Metabolism and nutrition disorders) | 19/291 | 16/255 | 30/449
Hyperlipidaemia (Metabolism and nutrition disorders) | 31/291 | 9/255 | 7/449
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 23/291 | 15/255 | 13/449
Arthralgia (Musculoskeletal and connective tissue disorders) | 47/291 | 20/255 | 29/449
Back pain (Musculoskeletal and connective tissue disorders) | 43/291 | 23/255 | 30/449
Muscle spasms (Musculoskeletal and connective tissue disorders) | 25/291 | 16/255 | 22/449
Myalgia (Musculoskeletal and connective tissue disorders) | 32/291 | 18/255 | 19/449
Pain in extremity (Musculoskeletal and connective tissue disorders) | 41/291 | 15/255 | 16/449
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21/291 | 17/255 | 18/449
Dizziness (Nervous system disorders) | 30/291 | 16/255 | 26/449
Headache (Nervous system disorders) | 73/291 | 34/255 | 53/449
Hypoaesthesia (Nervous system disorders) | 19/291 | 12/255 | 4/449
Neuropathy peripheral (Nervous system disorders) | 34/291 | 8/255 | 24/449
Paraesthesia (Nervous system disorders) | 17/291 | 11/255 | 10/449
Anxiety (Psychiatric disorders) | 27/291 | 6/255 | 22/449
Depression (Psychiatric disorders) | 50/291 | 32/255 | 30/449
Insomnia (Psychiatric disorders) | 46/291 | 27/255 | 31/449
Erectile dysfunction (Reproductive system and breast disorders) | 24/291 | 11/255 | 10/449
Cough (Respiratory, thoracic and mediastinal disorders) | 45/291 | 46/255 | 53/449
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21/291 | 12/255 | 10/449
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 20/291 | 7/255 | 9/449
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 27/291 | 15/255 | 20/449
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 18/291 | 7/255 | 9/449
Night sweats (Skin and subcutaneous tissue disorders) | 15/291 | 12/255 | 17/449
Pruritus (Skin and subcutaneous tissue disorders) | 24/291 | 17/255 | 16/449
Rash (Skin and subcutaneous tissue disorders) | 44/291 | 25/255 | 29/449
Hypertension (Vascular disorders) | 27/291 | 5/255 | 8/449

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.